CLINICAL TRIAL: NCT00064077
Title: A Randomized Phase III Trial Of Paclitaxel Plus Cisplatin Versus Vinorelbine Plus Cisplatin Versus Gemcitabine Plus Cisplatin Versus Topotecan Plus Cisplatin In Stage IVB, Recurrent Or Persistent Carcinoma of the Cervix
Brief Title: Comparison of Four Combination Chemotherapy Regimens Using Cisplatin in Treating Patients With Stage IVB, Recurrent, or Persistent Cancer of the Cervix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0204; NCI-2012-02540 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000306463; GOG-0204 (Other: Gynecologic Oncology Group); GOG-0204 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-08

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Recurrent Cervical Carcinoma; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Paclitaxel; Taxes; Topotecan; Vinorelbine

ARMS (4):
- Arm I (paclitaxel, cisplatin) (Experimental): Patients receive paclitaxel IV over 24 hours on day 1 and cisplatin IV over 1-4 hours on day 2.
  Interventions: Drug: Cisplatin; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm II (vinorelbine, cisplatin) (Experimental): Patients receive vinorelbine IV over 6-10 minutes on days 1 and 8 and cisplatin IV over 1-4 hours on day 1.
  Interventions: Drug: Cisplatin; Other: Quality-of-Life Assessment; Drug: Vinorelbine Tartrate
- Arm III (gemcitabine, cisplatin) (Experimental): Patients receive gemcitabine IV over 30-60 minutes on days 1 and 8 and cisplatin as in arm II.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Other: Quality-of-Life Assessment
- Arm IV (topotecan, cisplatin) (Experimental): Patients receive topotecan IV over 30 minutes on days 1-3 and cisplatin as in arm II.
  Interventions: Drug: Cisplatin; Other: Quality-of-Life Assessment; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
  Arms: Arm III (gemcitabine, cisplatin)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (paclitaxel, cisplatin)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Arm IV (topotecan, cisplatin)
Drug: Vinorelbine Tartrate — Given IV
  Other Names: Biovelbin; Eunades; KW-2307; Navelbine; Navelbine Ditartrate; NVB; Vinorelbine Ditartrate
  Arms: Arm II (vinorelbine, cisplatin)

SUMMARY:
This randomized phase III trial is studying four combination chemotherapy regimens using cisplatin to compare how well they work in treating women with stage IVB, recurrent, or persistent cancer of the cervix. Drugs used in chemotherapy such as cisplatin, paclitaxel, vinorelbine, gemcitabine, and topotecan, use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen containing cisplatin is most effective in treating cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the survival and response of patients with stage IVB, recurrent, or persistent carcinoma of the cervix when treated with paclitaxel and cisplatin vs vinorelbine and cisplatin vs gemcitabine and cisplatin vs topotecan and cisplatin.

II. Compare the toxic effects of these regimens in these patients. III. Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive paclitaxel IV over 24 hours on day 1 and cisplatin IV over 1-4 hours on day 2.

ARM II: Patients receive vinorelbine IV over 6-10 minutes on days 1 and 8 and cisplatin IV over 1-4 hours on day 1.

ARM III: Patients receive gemcitabine IV over 30-60 minutes on days 1 and 8 and cisplatin as in arm II.

ARM IV: Patients receive topotecan IV over 30 minutes on days 1-3 and cisplatin as in arm II.

In all arms, treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before courses 2 and 5, and at 9 months after study entry.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix

  * Stage IVB, recurrent, or persistent disease
* Not amenable to curative surgery and/or radiotherapy
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by palpation, plain x-ray, CT scan, or MRI OR at least 10 mm by spiral CT scan
  * Biopsy confirmation required if lesion is less than 30 mm
  * Target lesion must be outside of a previously irradiated field
* No craniospinal metastases
* Performance status - GOG 0-1
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times normal
* Alkaline phosphatase no greater than 3 times normal
* AST no greater than 3 times normal
* Creatinine ≤ 1.2 mg/dL
* Creatinine > 1.2 mg/dL but < 1.5 mg/dL AND creatinine clearance ≥ 50 mL/min
* No bilateral hydronephrosis not alleviated by ureteral stents or percutaneous drainage
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior or concurrent malignancy within the past 5 years except nonmelanoma skin cancer
* No prior malignancy whose treatment contraindicates the current study therapy
* No concurrent clinically significant infection
* No concurrent cytokines
* At least 6 weeks since prior chemoradiotherapy and recovered
* No prior chemotherapy (except when concurrently administered with radiotherapy)
* At least 3 weeks since prior radiotherapy and recovered
* Recovered from prior surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2003-05; Primary Completion 2011-01 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Monk, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2003 through April 2007, 513 patients were enrolled. Interim analysis recommended early closure for futility in January 2004.
Pre-assignment Details: Until January 2004, the study consisted of only two arms. Interim analysis recommended early closure for futility. 41 patients were enrolled until that point. These 41 patients were excluded from analysis. Two more arms were added and the study re-opened with 4 arms. The 472 patients enrolled after 1/26/2004 were included in analysis.
Groups:
- Arm III (Gemcitabine, Cisplatin): Patients receive gemcitabine IV over 30-60 minutes on days 1 and 8 and cisplatin as in arm II.
  Cisplatin: Given IV
  Gemcitabine Hydrochloride
  Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin)
Started | 118 | 117 | 119 | 118
Completed | 103 (Evaluable (treatment)) | 108 (Evaluable (treatment)) | 112 (Evaluable (treatment)) | 111 (Evaluable (treatment))
Not Completed | 15 | 9 | 7 | 7
Not completed — Improper prior treatment | 1 | 0 | 0 | 0
Not completed — Poor risk | 2 | 0 | 1 | 1
Not completed — Pathology | 10 | 7 | 3 | 4
Not completed — No surgery | 0 | 0 | 1 | 0
Not completed — No tumor | 0 | 0 | 1 | 0
Not completed — Other reasons | 2 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Evaluable (treatment)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin) | Total
Number analyzed (Participants) | 103 | 108 | 112 | 111 | 434
Age, Continuous [Median (Full Range); unit: years] | 50 [29 to 81] | 49 [24 to 76] | 45 [20 to 89] | 48 [25 to 75] | 48 [20 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 108 | 112 | 111 | 434
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 10 | 20 | 19 | 65
  Not Hispanic or Latino | 75 | 90 | 86 | 78 | 329
  Unknown or Not Reported | 12 | 8 | 6 | 14 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 1 | 5
  Asian | 4 | 6 | 3 | 4 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 20 | 23 | 17 | 79
  White | 75 | 79 | 80 | 82 | 316
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Duration of Overall Survival (OS)
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Baseline, every other cycle during treatment, then every 3 months for 2 years, the every 6 months for 3 years (up to 5 years)
Population: Evaluable (treatment)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin)
Number analyzed (Participants) | 103 | 108 | 112 | 111
months | 12.87 [10.02 to 16.76] | 9.99 [8.25 to 12.25] | 10.28 [7.62 to 11.60] | 10.25 [8.61 to 11.66]

2. Secondary Outcome: Frequency of Response Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above.
Time Frame: as for outcome 1
Population: Evaluable (treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin)
Number analyzed (Participants) | 103 | 108 | 112 | 111
Participants
  Complete Response | 3 | 8 | 1 | 2
  Partial Response | 27 | 20 | 24 | 24
  Stable Disease | 50 | 46 | 54 | 53
  Progressive Disease/other | 23 | 34 | 33 | 32

3. Secondary Outcome: Duration of Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 1
Population: Evaluable (treatment)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin)
Number analyzed (Participants) | 103 | 108 | 112 | 111
months | 5.82 [4.53 to 7.59] | 3.98 [3.19 to 5.16] | 4.70 [3.58 to 5.59] | 4.57 [3.71 to 5.75]

4. Secondary Outcome: Patient-reported Quality of Life as Measured by the Functional Assessment of Cancer Therapy (FACT)-Cervical Trial Outcome of Index (FACT-Cx TOI)
Description: The FACT-Cx TOI is a scale for assessing general QOL of cervical cancer patients.consisting of three subscales: Physical Well Being (7 items), Functional Well Being (7 items), and Cervical Cancer subscale (15 items). Each item in the FACT-Cx TOI was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative statements (or questions), reversal was performed prior to score calculation. According to the FACIT measurement system, a subscale score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the subscale. The score is calculated as the sum of the subscale scores if more than 80% of the FACT-Cx TOI items provide valid answers and all of the component subscales have valid scores. The score ranges 0-116 with a large score suggesting better QOL.
Time Frame: Baseline (pre-cycle 1), Pre-cycle 2, Pre-cycle 5, 9 months post cycle 1
Population: Patients who provided baseline and ≥ one follow-up assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin)
Number analyzed (Participants) | 86 | 89 | 92 | 96
units on a scale
  Baseline | 66.6 (17.6) | 69.1 (18.6) | 67.9 (19.5) | 68.1 (19.2)
  Pre-cycle 2 | 65.2 (17.6) | 65.5 (15.8) | 65.3 (18.2) | 66.2 (16.3)
  Pre-cycle 5 | 70.5 (16.5) | 66.6 (17.4) | 64.5 (16.5) | 68.4 (15.5)
  9 months post cycle 1 | 71.9 (16.6) | 69.9 (18.8) | 68.6 (19.5) | 70.9 (17.9)

5. Secondary Outcome: Pain, Assessed by Brief Pain Inventory
Description: Single item from the Brief Pain Inventory (BPI) assessing "worst pain" in the past 24 hours, on a 0-10 scale with a higher score indicating more pain than a low score.
Time Frame: Baseline (pre-cycle 1), Pre-cycle 2, Pre-cycle 5, 9 months post cycle 1
Population: Patients who provided baseline and ≥ one follow-up assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin)
Number analyzed (Participants) | 74 | 83 | 86 | 92
units on a scale
  Baseline | 4.0 (2.8) | 3.9 (3.2) | 3.3 (3.0) | 3.6 (3.3)
  Pre-cycle 2 | 3.5 (2.9) | 3.5 (2.8) | 3.4 (3.0) | 3.6 (3.1)
  Pre-cycle 5 | 3.6 (3.1) | 4.0 (2.7) | 3.5 (3.0) | 2.5 (3.0)
  9 months post cycle 1 | 2.3 (3.0) | 3.2 (2.9) | 3.7 (3.0) | 2.9 (2.7)

6. Secondary Outcome: Patient Reported Neurotoxicity Symptoms as Measured With the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity Subscale (Short Version) (FACT/GOG-Ntx Subscale).
Description: The FACT/GOG-Ntx subscale contains 4 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative items, reversal was performed prior to score calculation. According to the FACIT measurement system, the Ntx score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the scale. The Ntx score ranges 0-16 with a large score suggests less neurotoxicity.
Time Frame: Baseline (pre-cycle 1), Pre-cycle 2, Pre-cycle 5, 9 months post cycle 1
Population: Patients who provided baseline and ≥ one follow-up assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin)
Number analyzed (Participants) | 84 | 89 | 91 | 96
units on a scale
  Baseline | 14.4 (2.9) | 13.5 (3.4) | 14.2 (2.9) | 14.1 (3.5)
  Pre-cycle 2 | 14.1 (3.2) | 13.3 (3.6) | 13.7 (3.5) | 14.2 (3.2)
  Pre-cycle 5 | 13.1 (3.5) | 13.1 (3.7) | 14.1 (3.0) | 14.4 (3.2)
  9 months post cycle 1 | 11.1 (5.2) | 11.4 (4.7) | 12.3 (3.7) | 13.1 (3.5)

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment , and up to 5 years in follow-up.
Arm/Group | Arm I (Paclitaxel, Cisplatin) | Arm II (Vinorelbine, Cisplatin) | Arm III (Gemcitabine, Cisplatin) | Arm IV (Topotecan, Cisplatin)
Serious Adverse Events (participants affected / at risk) | 42/103 | 39/108 | 38/112 | 38/111
Other Adverse Events (participants affected / at risk) | 101/103 | 105/108 | 109/112 | 108/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Cisplatin) (N=103) | Arm II (Vinorelbine, Cisplatin) (N=108) | Arm III (Gemcitabine, Cisplatin) (N=112) | Arm IV (Topotecan, Cisplatin) (N=111)
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 2
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 8 | 2 | 7
Transfusion Prbc's (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Thrombosis Embolism (Cardiac disorders) | 5 | 9 | 5 | 3
Ischemia/Cardiac Infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac Left Ventricular Function (Cardiac disorders) | 0 | 0 | 0 | 1
Hypotension (Cardiac disorders) | 1 | 2 | 1 | 0
Other Cardiovascular (Cardiac disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 0
Diarrhea Without Colostomy (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Dehydration (Gastrointestinal disorders) | 5 | 2 | 3 | 1
Anorexia (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fistula Rectal/Anal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea With Colostomy (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fistula Intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gi Other (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Fever(No Neutropenia) (General disorders) | 0 | 2 | 2 | 0
Bone Pain (General disorders) | 0 | 0 | 1 | 1
Abdominal Pain (General disorders) | 3 | 2 | 1 | 3
Pain Rectal/Perirectal (General disorders) | 1 | 0 | 0 | 0
Pain Other (General disorders) | 1 | 2 | 1 | 1
Allergic Reaction (Immune system disorders) | 2 | 0 | 0 | 0
Febrile With Neutropenia (Infections and infestations) | 6 | 2 | 2 | 2
Infection Without Neutropenia (Infections and infestations) | 7 | 4 | 4 | 5
Infection With Grade 3/4 Neutropenia (Infections and infestations) | 1 | 2 | 0 | 3
Infection No Anc (Infections and infestations) | 1 | 0 | 0 | 1
Catheter-Related Infection (Infections and infestations) | 0 | 0 | 1 | 0
Infection Other (Infections and infestations) | 0 | 1 | 0 | 0
Other Infection (Infections and infestations) | 0 | 3 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic Other (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Ataxia(Incoordination) (Nervous system disorders) | 1 | 0 | 0 | 0
Cns Cerebrovascular Ischemia (Nervous system disorders) | 1 | 0 | 0 | 0
Speech Impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Creatinine (Renal and urinary disorders) | 1 | 2 | 2 | 1
Renal Failure (Renal and urinary disorders) | 1 | 2 | 0 | 0
Fistula (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureteral Obstruction (Renal and urinary disorders) | 1 | 2 | 4 | 4
Renal/Gu Other (Renal and urinary disorders) | 1 | 0 | 0 | 0
Other Genitourinary/Renal (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wound Infectious (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Prothrombin Time (Vascular disorders) | 0 | 0 | 0 | 1
Hemorrhage With Grade 3/4 Thrombocytopenia (Vascular disorders) | 0 | 0 | 1 | 0
Melena/Gi Bleeding (Vascular disorders) | 1 | 0 | 1 | 1
Vaginal Bleeding (Vascular disorders) | 0 | 1 | 2 | 3
Hemoptysis (Vascular disorders) | 0 | 0 | 1 | 0
Rectal Bleeding/Hematochezia (Vascular disorders) | 0 | 0 | 1 | 0
Other Hemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Cisplatin) (N=103) | Arm II (Vinorelbine, Cisplatin) (N=108) | Arm III (Gemcitabine, Cisplatin) (N=112) | Arm IV (Topotecan, Cisplatin) (N=111)
Leukopenia (Blood and lymphatic system disorders) | 92 | 98 | 90 | 102
Anemia (Blood and lymphatic system disorders) | 94 | 100 | 104 | 106
Thrombocytopenia (Blood and lymphatic system disorders) | 36 | 32 | 88 | 87
Neutropenia (Blood and lymphatic system disorders) | 92 | 94 | 76 | 102
Otherhematologic (Blood and lymphatic system disorders) | 38 | 53 | 57 | 57
Lymphatics (Blood and lymphatic system disorders) | 1 | 3 | 2 | 5
Thrombosis Embolism (Cardiac disorders) | 5 | 7 | 2 | 5
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Left Ventricular Function (Cardiac disorders) | 1 | 0 | 1 | 2
Other Cardiovascular (Cardiac disorders) | 22 | 15 | 11 | 13
Inner Ear/Hearing (Ear and labyrinth disorders) | 10 | 14 | 17 | 11
Other Hearing (Ear and labyrinth disorders) | 2 | 1 | 2 | 2
Endocrine (Endocrine disorders) | 9 | 4 | 4 | 5
Ocular (Eye disorders) | 6 | 5 | 4 | 8
Nausea (Gastrointestinal disorders) | 62 | 64 | 59 | 61
Vomiting (Gastrointestinal disorders) | 59 | 51 | 57 | 49
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 18 | 10 | 21 | 13
Other Gastrointestinal (Gastrointestinal disorders) | 65 | 67 | 75 | 66
Fatigue (General disorders) | 74 | 82 | 90 | 85
Other Constitutional (General disorders) | 17 | 23 | 27 | 28
Myalgia (General disorders) | 19 | 9 | 13 | 12
Other Pain (General disorders) | 33 | 47 | 40 | 40
Hepatic (Hepatobiliary disorders) | 17 | 13 | 16 | 20
Allergic Reaction (Immune system disorders) | 10 | 6 | 4 | 9
Other Allergy (Immune system disorders) | 1 | 4 | 3 | 3
Febrile With Neutropenia (Infections and infestations) | 13 | 15 | 6 | 11
Infection Without Neutropenia (Infections and infestations) | 19 | 12 | 19 | 9
Other Infection (Infections and infestations) | 11 | 12 | 5 | 13
Metabolic (Metabolism and nutrition disorders) | 50 | 50 | 49 | 48
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 | 6 | 9 | 8
Neuropathy Sensor (Nervous system disorders) | 37 | 33 | 21 | 23
Otherneurologic (Nervous system disorders) | 27 | 30 | 28 | 22
Creatinine (Renal and urinary disorders) | 15 | 18 | 20 | 16
Other Genitourinary/Renal (Renal and urinary disorders) | 10 | 9 | 6 | 14
Sexual/Reproductive (Reproductive system and breast disorders) | 0 | 0 | 2 | 2
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 20 | 16 | 11 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 65 | 26 | 22 | 48
Rash Desquamation (Skin and subcutaneous tissue disorders) | 5 | 3 | 7 | 7
Other Dermatologic (Skin and subcutaneous tissue disorders) | 15 | 14 | 11 | 7
Coagulation (Vascular disorders) | 0 | 3 | 1 | 1
Hemorrhage (Vascular disorders) | 6 | 7 | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less